CLINICAL TRIAL: NCT00641940
Title: Girls in Transition Study: Helping Girls Enter the Teenage Years
Acronym: GT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Swarthmore College (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Jane E. Gillham, Ph.D., Swarthmore College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 803680
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2008-03-24 (Estimated); Status verified 2008-03

CONDITIONS: Depression; Anxiety
Keywords: Prevention; Girls; Resilience
MeSH Terms: conditions — Depression; Anxiety Disorders

ARMS (2):
- 1 (Experimental): Girls in Transition (GT) program
  Interventions: Behavioral: Girls in Transition (GT) program
- 2 (Other): Waitlist control
  Interventions: Behavioral: Waitlist Control

INTERVENTIONS:
Behavioral: Girls in Transition (GT) program — In the 11-session after-school GT program, girls learn cognitive and behavioral skills related to intrapersonal, interpersonal, and social/contextual risk factors for depression.
  Other Names: GT #1
  Arms: 1
Behavioral: Waitlist Control — Participants in the waitlist control group will complete the GT program during the third year of the study.
  Other Names: GT #2
  Arms: 2

SUMMARY:
This is a pilot study of the Girls in Transition (GT) program, an intervention designed to promote resilience and reduce gender-related risk factors for depression. The goal of the study is to gather preliminary data on the effects of the GT program.

DETAILED DESCRIPTION:
Gender differences in rates of depression emerge during adolescence. Although rates of depression increase for both boys and girls during adolescence, the increase is more dramatic for girls. By late adolescence, girls are twice as likely as boys to develop depression. Because the transition to adolescence has been identified as a period of increased risk for girls, preventive interventions targeting early adolescent girls may promote resilience and prevent depression. The Girls in Transition (GT) program is a group intervention for 6th through 8th grade girls and is designed to address risk factors that are specific to girls. This study evaluates the effectiveness of the GT intervention in promoting coping strategies, preventing symptoms of depression and anxiety, and providing benefits in other outcomes related to depression, such as self-image.

Adolescents in this study will be assigned to one of two conditions: a group that will participate in the GT program in Spring 2006 (GT #1), or a waitlist control group that will participate in the GT program approximately two years later (GT #2). Students who participate in the program will attend eleven 90-minute after-school sessions led by the investigators. In the GT program, students learn cognitive-behavioral skills (such as strategies to cope with emotions and negative thinking) and problem-solving skills (such as assertiveness), and they discuss societal messages about women's appearance and roles. Adolescent participants will complete questionnaires about coping strategies, self-image, and feelings of hopelessness, depression and anxiety at five points during the study: at the beginning of the study (baseline) and at follow-ups approximately 6, 12, 16, and 24 months after baseline. In addition, students will complete an interview at baseline and then again 12 months later about experiences in which they have coped with stressful situations. Parents will complete a questionnaire about their child's life events at three assessment points (baseline and at follow-ups approximately 12 and 24 months after baseline).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Student in grades 6 through 8
* Student in participating school

Exclusion Criteria:

* Male

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Adolescents' coping strategies by self-report | Measured at baseline and follow-ups approximately 6, 12, and 24 months after baseline
Adolescents' depressive symptoms by self-report | Measured at baseline and follow-ups approximately 6, 12, 16, and 24 months after baseline

SECONDARY OUTCOMES:
Adolescents' symptoms of anxiety by self-report | Measured at baseline and follow-ups approximately 6, 12, 16, and 24 months after baseline
Adolescents' feelings of hopelessness by self-report | Measured at baseline and follow-ups approximately 6, 12, and 24 months after baseline
Adolescents' perceptions of their physical appearance by self-report | Measured at baseline and follow-ups approximately 6, 12, and 24 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jane E. Gillham, Ph.D., Principal Investigator — Swarthmore College
Locations (1):
- Swarthmore College, Swarthmore, Pennsylvania, United States